CLINICAL TRIAL: NCT04488653
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Determine the Safety and Efficacy of Oligopin® on Metabolic Risk Factors in Subjects With Metabolic Syndrome
Brief Title: A Study to Determine the Safety and Efficacy of Oligopin® on Metabolic Risk Factors in Subjects With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Les Derives Resiniques et Terpeniques (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19PMHD
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Oligopin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligopin® (Experimental): Oligopin® contains French Maritime Pine Bark Extract
  Interventions: Dietary Supplement: Oligopin®
- Placebo (Placebo Comparator): Placebo is a mixture of different inert compounds
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligopin® — French Maritime Pine Bark Extract - 100mg/day
  Arms: Oligopin®
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The safety and efficacy of Oligopin® will be compared against a placebo to evaluate the effect on metabolic risk factors in subjects with metabolic syndrome. During the 84-day study period it is hypothesized that HDL cholesterol will increase and systolic blood pressure will decrease therefore lowering CVD risk factors after supplementation with Oligopin®. Additionally, it is hypothesized that Oligopin® supplementation will reduce fasting glucose levels.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a combination of risk factors for chronic conditions such as cardiovascular disease (CVD) and type 2 diabetes (T2D). These risk factors include obesity (particularly abdominal obesity), high blood pressure, elevated triglycerides, low high-density lipoprotein (HDL) cholesterol, and elevated fasting blood glucose. MetS reflects overnutrition and sedentary lifestyles as the prevalence of MetS increases concomitantly with these lifestyle choices. Most recent estimates suggest that approximately 19.1% of the Canadian population, 34.2% of the US population, and 24.3% of the European population have MetS. Significantly, the prevalence of MetS in adults aged 18-39 has increased dramatically over the last 2 decades.

MetS commonly precedes the development of CVD and is associated with a 2-fold increase in the risk of CVD mortality. MetS also increases the risk of developing T2D and is suggested to be extremely prevalent (90-95%) in Caucasian individuals diagnosed with T2D. Indeed, the presence of even one MetS risk factor early in life increases the chances of developing a chronic disease later in life. Currently, MetS risk factors are estimated to be present in 4.8-7% of individuals from 18 to 30 years of age. Therefore, preventing the development of or treating these risk factors earlier in life could reduce the development of chronic disease.

The pathogenic mechanisms of MetS remain to be fully elucidated, however insulin resistance (IR) appears to play a pivotal role in the initiation and progression of the syndrome. Abdominal obesity is a well-known contributor to IR. Abdominal fat accumulation increases the supply of free fatty acids (FFAs) to the liver and indirectly results in an increase in plasma low-density lipoprotein (LDL) cholesterol and a decrease in HDL cholesterol. IR also elevates fasting blood glucose levels due to the suppression of hepatic glycogen synthesis and impairs postprandial glucose control by reducing insulin stimulated glucose uptake by peripheral tissues.

There is a need for natural interventions that aid in the prevention and treatment of MetS risk factors as the prevalence of overnutrition and sedentary lifestyles continues to increase. This study will assess the ability of Oligopin® to improve abdominal obesity, fasting blood glucose, postprandial glucose and insulin response, and HDL-cholesterol levels as these outcomes reliably predict an individual's MetS risk. Oligopin® is a French Maritime Pine Bark Extract (FMPBE) obtained from the pine tree Pinus pinaster. It is rich in low molecular weight oligomeric procyanidins (OPC) with 20% of OPCs in the form of dimers as compared to the most studied FMPBE Pycogenol®, which contains only 5% of OPCs as dimers.

Recently, Oligopin® supplementation was shown to reduce CVD risk factors. In a randomized, double-blind, placebo-controlled clinical trial, Oligopin® consumption increased HDL cholesterol levels and reduced systolic blood pressure and oxidized LDL (oxLDL) levels in stage 1 hypertensive individuals. This is significant as low HDL was reported to be the most prevalent risk factor for the development of MetS in young adults. FMPBE supplementation has also been shown to reduce fasting glucose levels in individuals with T2D. Interestingly, FMPBE is a potent inhibitor of α-glucosidase, which catalyses the breakdown of oligosaccharides in the small intestine to permit glucose resorption. Therefore, it is possible that Oligopin® may reduce fasting glucose levels and control postprandial hyperglycemia. This randomized, double-blind, placebo-controlled study will determine the efficacy of Oligopin® to improve markers of metabolic risk in subjects with MetS.

ELIGIBILITY:
Inclusion Criteria:

* Provided voluntary, written, informed consent to participate in the study
* Males and females between 18 and 55 years of age, inclusive
* Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-
* Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner at least 6 months prior to screening
* BMI between 25 to 34.9 kg/m2, inclusive
* Subjects with three or more of the following markers associated with metabolic syndrome:
* Abdominal obesity: waist circumference > 102 cm (40 inches) in men and > 88 cm (35 inches) in women
* Hypertension: systolic blood pressure > 130 mmHg or diastolic blood pressure > 85 mmHg
* Elevated fasting glucose > 5.6 mmol/L (> 100 mg/dL) and < 7.0 mmol/L (< 126 mg/dL) and/or elevated HbA1c (6.0-6.4%)
* Elevated TG: > 150 mg/dL (1.7 mmol/L)
* Low HDL-C: < 40 mg/dL (1.03 mmol/L) in men and < 50 mg/dL (1.29 mmol/L) in women
* Stable weight defined as < 5% change in body weight in six months prior to beginning of study
* Agrees to maintain current diet and exercise routine during the study
* Agrees to comply with all study-related procedures
* Otherwise healthy as determined by medical history, laboratory results, and physical exam as assessed by the Qualified Investigator (QI)

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the trial
* Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
* Participation in other clinical research trials 30 days prior to screening
* Individuals who are unable to give informed consent
* Current or history of any significant diseases of the gastrointestinal tract that may impact study outcomes as assessed by the QI
* Unstable metabolic disease or chronic diseases as assessed by the QI
* Unstable hypertension as assessed by the QI
* Type I or Type II diabetes
* Individuals with hypercholesterolemia and/or elevated triglycerides who are receiving medications to modulate lipid metabolism, as in Sections 6.3.1 and 6.3.2
* Individuals with an autoimmune disease or who are immune-compromised
* Self-reported HIV-, Hepatitis B- and/or C-positive diagnosis
* History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom free for 6 months
* Self-reported current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
* Self-reported medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
* Self-reported blood/bleeding disorder
* Serious cardiovascular or respiratory disease as assessed by the QI.
* Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
* Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
* Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients, or the ingredients in the test meal
* Current use of prescribed medications listed in Section 6.3.1
* Current use of over-the-counter medications, supplements, foods and/or drinks listed in Section 6.3.2
* Medical use of cannabinoid products
* Chronic recreational use of cannabinoid products (>2 times/week). Occasional use will be assessed by the QI on a case-by-case basis
* Use of tobacco or nicotine-containing products within 60 days of screening
* Alcohol or drug abuse within the last 12 months
* High alcohol intake (average of >2 standard drinks per day
* Clinically significant abnormal laboratory results at screening as assessed by the QI
* Any other condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-10-19 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Fasting blood sugar level | 84 days
  Change in fasting blood sugar from baseline to day 84 between Oligopin® and placebo.

SECONDARY OUTCOMES:
Fasting insulin concentration | Baseline, day 42 and day 84
  Change in fasting insulin between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Fasting glucose level | Baseline, day 42 and day 84
  Change in fasting glucose between Oligopin® and placebo baseline to day 42, baseline to day 84, and from day 42 to day 84
Concentration of fasting low-density lipoprotein (LDL) | Baseline, day 42 and day 84
  Change in fasting LDL between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Change in fasting oxidized LDL (oxLDL). | Baseline, day 42 and day 84
  Change in fasting oxLDL between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Change in fasting high-density lipoprotein (HDL) | Baseline, day 42 and day 84
  Change in fasting HDL between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Change in fasting total cholesterol | Baseline, day 42 and day 84
  Change in fasting total cholesterol between Oligopin® and placebo baseline to day 42, baseline to day 84, and from day 42 to day 84
Postprandial glucose at 20, 30, 90, or 120 min after meal | Baseline, day 42 and day 84
  Change in postprandial glucose between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Postprandial insulin at 20, 30, 90, or 120 min after meal | Baseline, day 42 and day 84
  Change in postprandial glucose between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
BMI | Baseline, day 42 and day 84
  Change in BMI between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Waist circumference | Baseline, day 42 and day 84
  Change in waist circumference between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Blood pressure | Baseline, day 42 and day 84
  Change in systolic and diastolic blood pressure between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Heart rate | 84 days
  Change in heart rate between Oligopin® and placebo from baseline to day 42, baseline to day 84, and from day 42 to day 84
Alanine aminotransferase (ALT) | Pre-baseline and 84 days
  Change in ALT between Oligopin® and placebo pre-baseline and day 84.
Aspartate transaminase (AST) | Pre-baseline and 84 days
  Change in AST between Oligopin® and placebo pre-baseline and day 84.
Total bilirubin | Pre-baseline and 84 days
  Change in total bilirubin between Oligopin® and placebo pre-baseline and day 84.
Creatinine | Pre-baseline and 84 days
  Change in creatinine between Oligopin® and placebo pre-baseline and day 84.
Sodium ion | Pre-baseline and 84 days
  Change in sodium ion between Oligopin® and placebo pre-baseline and day 84.
Potassium ion | Pre-baseline and 84 days
  Change in potassium ion between Oligopin® and placebo pre-baseline and day 84.
Chloride ion | Pre-baseline and 84 days
  Change in chloride ion between Oligopin® and placebo pre-baseline and day 84.
estimated glomerular filtration rate (eGFR) | Pre-baseline and 84 days
  Change in eGFR between Oligopin® and placebo pre-baseline and day 84.
White blood cell (WBC) count | Pre-baseline and 84 days
  Change in WBC count between Oligopin® and placebo pre-baseline and day 84.
Neutrophils | Pre-baseline and 84 days
  Change in neutrophil count between Oligopin® and placebo pre-baseline and day 84.
Lymphocytes | Pre-baseline and 84 days
  Change in lymphocyte count between Oligopin® and placebo pre-baseline and day 84.
Monocytes | Pre-baseline and 84 days
  Change in monocyte count between Oligopin® and placebo pre-baseline and day 84.
Eosinophils | Pre-baseline and 84 days
  Change in eosinophil count between Oligopin® and placebo pre-baseline and day 84.
Basophils | Pre-baseline and 84 days
  Change in basophil count between Oligopin® and placebo pre-baseline and day 84.
Red blood cell (RBC) | Pre-baseline and 84 days
  Change in RBC count between Oligopin® and placebo pre-baseline and day 84.
Hemoglobin | Pre-baseline and 84 days
  Change in hemoglobin level between Oligopin® and placebo pre-baseline and day 84.
Hematocrit | Pre-baseline and 84 days
  Change in hematocrit level between Oligopin® and placebo pre-baseline and day 84.
Platelet | Pre-baseline and 84 days
  Change in platelet count between Oligopin® and placebo pre-baseline and day 84.
Mean corpuscular volume (MCV) | Pre-baseline and 84 days
  Change in MCV level between Oligopin® and placebo pre-baseline and day 84.
Mean corpuscular hemoglobin (MCH) | Pre-baseline and 84 days
  Change in MCH level between Oligopin® and placebo pre-baseline and day 84.
Mean corpuscular hemoglobin concentration (MCHC) | Pre-baseline and 84 days
  Change in MCHC level between Oligopin® and placebo pre-baseline and day 84.
Mean platelet volume (MPV) | Pre-baseline and 84 days
  Change in MPV level between Oligopin® and placebo pre-baseline and day 84.
Red cell distribution width (RDW) | Pre-baseline and 84 days
  Change in RDW level between Oligopin® and placebo pre-baseline and day 84.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No